CLINICAL TRIAL: NCT03920995
Title: Creation of a Multi-center Database Registry to Study Real World Thalamus Volume Changes by Use of Artificial Intelligence in Patients With Multiple Sclerosis (MS)
Brief Title: Multi-center Database Registry to Study Thalamus Changes Using AI in MS
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director and Professor, University at Buffalo
Other Study IDs: N/A-NI-MS-PI-13632
Record Dates: First submitted 2019-03-12; First posted 2019-04-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the Investigator's propose to validate a newly developed approach, DeepGRAI (Deep Gray Rating via Artificial Intelligence), to simplify the calculation of thalamic atrophy in a clinical routine and allow academic and community neurologists to plan, perform, and publish novel and influential clinical research using data from clinical routine, by employing deep machine learning (DML) pattern recognition (PR) information through use of artificial intelligence (AI).

DETAILED DESCRIPTION:
This is a multicenter, observational, retrospective, cross-sectional and longitudinal population study of brain volume changes in MS patients. The retrospective electronic medical record (EMR) and brain MRI image data will be collected at participating MS centers and de-identified data will be integrated into a central research database. All the data to be integrated into the database has already been collected by physicians at the centers as part of their routine clinical practice and is thus non-interventional and retrospective in nature. This new approach will be compared to existing approaches of brain volume measurement that are currently widely available. This breakthrough approach would lead to potentially abandoning classis measurement of the specific brain volume structures and would be applicable in real-time in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with relapsing-remitting (RR) MS
2. Access to raw MRI index scan images that meet all of the below criteria

   1. MRI scan image acquired at index
   2. The scan was performed on 1.5T or 3T scanners
   3. The scan must have a T2-FLAIR sequence
3. Access to raw MRI post-index scan images that meet all of the below listed criteria

   1. MRI scan image acquired at post-index
   2. The scan was performed on 1.5T or 3T scanners
   3. The scan must have a T2-FLAIR sequence
4. Age 18-85 at index
5. Fulfilling the MRI scan and clinical data requirements outlined in Table 2
6. None of the exclusion criteria

Exclusion Criteria:

1. Have received an investigational drug or experimental procedure during the study period
2. Women who were pregnant, or lactating at index or during the post-index period
3. Patients who had a relapse 30 days prior to the selected MRI scan date
4. Patients who received steroid treatment 30 days prior to the selected MRI scan date
5. Presence of other neurologic diseases affecting CNS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Multiple sclerosis who have 2 MRI scans
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Multi-center registry of MRI scans | 2 years
  Measuring the ability of DeepGRAI to measure thalamus volume as a predictor of clinical outcomes for patients with multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No